CLINICAL TRIAL: NCT02540863
Title: Effectiveness of Myofascial Release and Exercises Therapy in the Treatment of Temporomandibular Disorders: a Randomized Clinical Trial
Brief Title: Miofascial Release and Exercises Therapy in the Treatment of Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, PhD (Lecturer), Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UAL-427
Record Dates: First submitted 2015-08-25; First posted 2015-09-04 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Temporomandibular Joint Disorders
Keywords: myofascial pain syndrome; exercise therapy; randomized controlled trial
MeSH Terms: conditions — Temporomandibular Joint Disorders; Myofascial Pain Syndromes | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- myofascial release protocol and Rocabado exercise therapy (Experimental): Myofascial Release Protocol:
  * Suboccipital release.
  * Compression - decompression of temporomandibular joint.
  * Horizontal release of temporomandibular joint.
  * Deep fascia release in temporal region.
  * Masseter deep fascia release.
  * Pterygoiddeep fascia release.
  * Intraoral pterygoid deep fascia release.
  Interventions: Other: myofascial release protocol and Rocabado exercise therapy
- exercise therapy (Active Comparator): Rocabado´s 6 x 6 exercises program utilizes six exercises six times by day. The patient is in supine position with a loop of 6 cm in the cervical area, and the therapist sits at the head of the bed.
  Interventions: Other: exercise therapy

INTERVENTIONS:
Other: myofascial release protocol and Rocabado exercise therapy
  Arms: myofascial release protocol and Rocabado exercise therapy
Other: exercise therapy
  Arms: exercise therapy

SUMMARY:
Objectives: The aim of this research is to compare the effectiveness of myofascial release therapy and exercise therapy on pain, quality of sleep, anxiety, trigger points, and joint sounds in individuals with temporomandibular disorders and myofascial pain-dysfunction syndrome.

Material and Methods: A single-blind randomized clinical trial will be conducted in a university research clinic. Sixty-four subjects with temporomandibular disorders and myofascial pain-dysfunction syndrome will be randomly assigned to physical therapy group (myofascial release protocol and Rocabado exercise therapy) and control group (exercise therapy). Intensity of pain, quality of life, quality of sleep, anxiety, trigger points, and joint sounds will be collected at baseline, and forty-eight hours after the intervention phase.

ELIGIBILITY:
Inclusion Criteria:

* Presence of myofascial pain with or without jaw opening limitation (Ia and Ib) according to the Research Diagnostic Criteria for Temporomandibular Disorders (RDC / TMD).
* A chief complaint of acute pain (duration < 6 months) in the temporomandibular joint on at least one side.
* The presence of joint clicking during jaw opening that was eliminated on protrusive opening.
* Agreement to attend evening therapy sessions.

Exclusion Criteria:

* Subjects with dental pain or tender muscles caused by systemic diseases.
* Major psychological disorders.
* A recent history of trauma in the face and neck area.
* Subjects wearing full or partial dentures.
* Edentulism.
* Therapeutic co-interventions during treatment.
* Indication for surgical treatment of temporomandibular joint.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Intensity of pain (100-mm VAS) | Changes from baseline in intensity of pain at twelve weeks
  A 100-mm VAS was used for determining pain intensity, ranging from 0 (no pain) to 100 (very severe pain).

SECONDARY OUTCOMES:
Quality of Sleep (Pittsburgh Sleep Quality Index - PSQI) | Changes from baseline in quality of sleep at twelve weeks
  PSQI was used to study the quality of sleep. It comprises 24 items where the individuals respond to 19 of these items, and individual living in the same dwelling (or hospital room) responds to remaining 5. Scores are obtained on each of 7 components of sleep quality: subjective quality, sleep latency, sleep duration, habitual sleep efficacy, sleep perturbations, use of hypnotic medication, and daily dysfunction. Each component is scored from 0 to 3 (0: no problems; 3: severe problems).
State and trait anxiety (state anxiety questionnaire and trait - STAI) | Changes from baseline in state and trait anxiety at twelve weeks
  Anxiety level were determined with the 40-item State-Trait Anxiety Inventory (STAI), which measures anxiety as a stable dimension of personality (trait or tendency to anxiety) and also includes a state subscale to detect anxiety behaviors. Subjects report their feelings in general for the trait scale and how they feel at the time of questionnaire completion for the state anxiety scale. The state anxiety scale indicates the feelings or sensations of anxiety (not at all, somewhat, moderately so, very much so) at a specific moment in time. The trait anxiety scale indicates the frequency with which anxiety is experienced (almost never, sometimes, often, almost, and always).
Physical parameters of active and passive mouth opening | Changes from baseline in active and passive mouth opening at twelve weeks
  The subjects were asked to open her/his mouth as much as possible for the measurement of active mouth opening without pain and maximal active mouth opening. Maximal passive mouth opening was measured after the application of downward pressure on the mandible by the second and third finger of the patient. The vertical overlap of the incisors was measured by a ruler (Helios-Preisser, Gammertingen, Germany) and recorded in mm for these parameters.
Physical parameters of pain in temporalis muscles | Changes from baseline in pain in temporalis muscles at twelve weeks
  Trigger points were assessed by palpation of temporal muscle (anterior, middle, and origin).
Physical parameters of lateral condyle pole and temporal tendon insertion pain | Changes from baseline in Lateral condyle pole and temporal tendon insertion pain at twelve weeks
  The muscles, tendon, and lateral condyles were palpated to the finger portion of the examiner´s finger applying a pressure on the muscle (1 Kg) and lateral condyles (0.5 Kg) being studied for 3-6s.
Physical parameters of clicking sound when opening / close palpation | Changes from baseline in clicking sound when opening / close palpation at twelve weeks
  Joint sounds during mouth opening and closing were assessed with the examiner's left index finger on the right joint and the right finger on pre-auricular area. The fingertip is placed anterior to the tragus of the ear. The patient is asked to slowly open as much as possible. After each closing, the subject must place the teeth in contact at a maximal intercuspal position. The patient open and close the mouth three times. Total number of sounds was recorded on both sides.
Physical parameters of pain in masseter muscles | Changes from baseline in pain in temporalis muscles at twelve weeks
  Trigger points were assessed by palpation of masseter muscle (anterior, deep, origin).
Physical parameters of pain in lateral pterygoid muscles | Changes from baseline in pain in lateral pterygoid muscles at twelve weeks
  Trigger points were assessed by palpation of lateral pterygoid muscle

REFERENCES:
- [Background] Hoffmann RG, Kotchen JM, Kotchen TA, Cowley T, Dasgupta M, Cowley AW Jr. Temporomandibular disorders and associated clinical comorbidities. Clin J Pain. 2011 Mar-Apr;27(3):268-74. doi: 10.1097/AJP.0b013e31820215f5. PMID 21178593
- [Background] Venancio Rde A, Camparis CM, Lizarelli Rde F. Low intensity laser therapy in the treatment of temporomandibular disorders: a double-blind study. J Oral Rehabil. 2005 Nov;32(11):800-7. doi: 10.1111/j.1365-2842.2005.01516.x. PMID 16202043
- [Background] Dworkin SF, LeResche L. Research diagnostic criteria for temporomandibular disorders: review, criteria, examinations and specifications, critique. J Craniomandib Disord. 1992 Fall;6(4):301-55. No abstract available. PMID 1298767
- [Background] Leblebici B, Pektas ZO, Ortancil O, Hurcan EC, Bagis S, Akman MN. Coexistence of fibromyalgia, temporomandibular disorder, and masticatory myofascial pain syndromes. Rheumatol Int. 2007 Apr;27(6):541-4. doi: 10.1007/s00296-006-0251-z. Epub 2006 Nov 10. PMID 17096090
- [Background] Manfredini D, Tognini F, Montagnani G, Bazzichi L, Bombardieri S, Bosco M. Comparison of masticatory dysfunction in temporomandibular disorders and fibromyalgia. Minerva Stomatol. 2004 Nov-Dec;53(11-12):641-50. English, Italian. PMID 15894939
- [Background] Aaron LA, Burke MM, Buchwald D. Overlapping conditions among patients with chronic fatigue syndrome, fibromyalgia, and temporomandibular disorder. Arch Intern Med. 2000 Jan 24;160(2):221-7. doi: 10.1001/archinte.160.2.221. PMID 10647761
- [Background] Balasubramaniam R, de Leeuw R, Zhu H, Nickerson RB, Okeson JP, Carlson CR. Prevalence of temporomandibular disorders in fibromyalgia and failed back syndrome patients: a blinded prospective comparison study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Aug;104(2):204-16. doi: 10.1016/j.tripleo.2007.01.012. Epub 2007 May 7. PMID 17482850
- [Background] Fraga BP, Santos EB, Farias Neto JP, Macieira JC, Quintans LJ Jr, Onofre AS, De Santana JM, Martins-Filho PR, Bonjardim LR. Signs and symptoms of temporomandibular dysfunction in fibromyalgic patients. J Craniofac Surg. 2012 Mar;23(2):615-8. doi: 10.1097/SCS.0b013e31824cd81a. PMID 22446432
- [Background] Rhodus NL, Fricton J, Carlson P, Messner R. Oral symptoms associated with fibromyalgia syndrome. J Rheumatol. 2003 Aug;30(8):1841-5. PMID 12913944
- [Background] Alonso-Blanco C, Fernandez-de-Las-Penas C, de-la-Llave-Rincon AI, Zarco-Moreno P, Galan-Del-Rio F, Svensson P. Characteristics of referred muscle pain to the head from active trigger points in women with myofascial temporomandibular pain and fibromyalgia syndrome. J Headache Pain. 2012 Nov;13(8):625-37. doi: 10.1007/s10194-012-0477-y. Epub 2012 Aug 31. PMID 22935970
- [Background] Nifosi F, Violato E, Pavan C, Sifari L, Novello G, Guarda Nardini L, Manfredini D, Semenzin M, Pavan L, Marini M. Psychopathology and clinical features in an Italian sample of patients with myofascial and temporomandibular joint pain: preliminary data. Int J Psychiatry Med. 2007;37(3):283-300. doi: 10.2190/PM.37.3.f. PMID 18314857
- [Background] Salvetti G, Manfredini D, Bazzichi L, Bosco M. Clinical features of the stomatognathic involvement in fibromyalgia syndrome: a comparison with temporomandibular disorders patients. Cranio. 2007 Apr;25(2):127-33. doi: 10.1179/crn.2007.019. PMID 17508633